CLINICAL TRIAL: NCT00768599
Title: A Multi-Center Randomized, Evaluator-Blinded, Vehicle Controlled, Parallel Group Comparison Study of the Safety and Efficacy of Econazole Nitrate Foam 1%, Econazole Nitrate 1% Cream, and Foam Vehicle in Subjects With Tinea Pedis
Brief Title: A Study of Econazole Foam 1% in Athlete's Foot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmDerma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D79-2902-07
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-12

CONDITIONS: Tinea Pedis; Athlete's Foot
Keywords: Econazole; Foam; Quinnova
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Econazole Nitrate Cream 1%
  Interventions: Drug: Econazole Nitrate Cream 1%
- 2 (Experimental): Econazole Nitrate Foam 1%
  Interventions: Drug: Econazole Nitrate Foam 1%
- 3 (Placebo Comparator): Vehicle Foam
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Econazole Nitrate Cream 1% — Topical cream, applied once daily for 4 weeks.
  Other Names: Econazole Nitrate Cream 1%, Fougera - Altana Inc.
  Arms: 1
Drug: Econazole Nitrate Foam 1% — Topical foam, applied once daily for 4 weeks.
  Other Names: Quinnova Econazole Nitrate Foam 1%
  Arms: 2
Drug: Vehicle Foam — Topical foam, applied once daily for 4 weeks.
  Other Names: Quinnova Foam Vehicle
  Arms: 3

SUMMARY:
This is a 6-week clinical study (4 weeks of treatment, once per day, plus a 2-week follow-up period) of a topical foam to treat athlete's foot. The active ingredient in the foam -- econazole nitrate 1% -- is the same active pharmaceutical ingredient in a cream that your doctor can currently prescribe to treat athlete's foot. This study will help to understand if the foam works the same as the cream to treat athlete's foot.

DETAILED DESCRIPTION:
Treating athlete's foot with a cream can leave a greasy, wet feeling on the foot that is uncomfortable to the user and messy on clothing and foot wear. A foam formulation that spreads easily and rubs-in easily that is as effective as the (reference) cream formulation in treating athlete's foot would be a benefit to the user. This study is designed to substantiate a clinical bridge between econazole nitrate foam 1% and econazole nitrate cream 1% based on clinical outcome, safety, and pharmacokinetic data. The study is (foam) vehicle-controlled and is randomized 1 to 1 to 1 (foam:cream:vehicle).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years or age and of either sex.
* Has a clinical diagnosis of tinea pedis with at least i) moderate scaling(interdigital and/or moccasin) and ii) mild erythema (interdigital only).
* Be willing to give informed consent.
* Be willing and able to give informed consent.
* Has microscopic evidence (positive KOH) of the presence of fungi. Evaluable subjects must have a positive KOH and a fungal culture positive for a dermatophyte at Baseline. Subjects with a positive KOH may be entered into the study pending the results of the fungal culture.
* Be in good health and free of any disease or physical condition which might, in the investigator's opinion, expose the subject to an unacceptable risk by study participation.
* Women of childbearing potential must have a negative urine pregnancy test and agree to use an effective, non-prohibited form of birth control for the duration of the study (abstinence, stabilized on oral contraceptives for at least two months, implant, injection, IUD, patch, NuvaRing, condom and spermicidal or diaphragm and spermicidal).

Exclusion Criteria:

* Is nursing or planning a pregnancy during the study.
* Has used topical antifungal or corticosteroid therapy or systemic antibacterial therapy within 30 days prior to the start of the study.
* Has received systemic antifungal therapy within 12 weeks prior to the start of the study medication.
* Has a history of diabetes mellitus or is immunocompromised (due to disease, e.g., HIV, or medications).
* Has concurrent tinea infection (in the opinion of the investigator). However, concurrent onychomycosis is allowed.
* Has any other skin disease which might interfere with the evaluation of tinea pedis.
* Is currently enrolled in an investigational drug or device study.
* Has received an investigational drug or treatment with an investigational device within 30 days prior to entering this study
* Is unreliable, including subjects with a history of drug or alcohol abuse.
* Has known hypersensitivity to any of the components of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Stacy Smith, MD, San Diego, California
  - Daniel Stewart, DO, Clinton Township, Michigan
  - Steven Kempers, MD, Fridley, Minnesota
  - Michael Gold, MD, Nashville, Tennessee
  - Michael Jarratt, MD, Austin, Texas
  - Leonard Swinyer, MD, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and ninety-eight (198) subjects were screened and 135 were enrolled/randomized in the study. Subjects with negative KOH evaluations in both regions (all scrapings negative) were considered Screen Failures and were not enrolled into the study. Subject enrollment and completion dates are March 27, 2008 - September 25, 2008.
Pre-assignment Details: Subjects who met the inclusion/exclusion criteria were randomized to receive Econazole Nitrate Foam 1%, Econazole Nitrate Cream 1%, or Foam vehicle in a 1:1:1 ratio.
Groups:
- Reference Drug: Econazole Nitrate Cream 1%
- Test Drug: Econazole Nitrate Foam 1%
- Control: Vehicle Foam
Period: Overall Study
Arm/Group | Reference Drug | Test Drug | Control
Started | 45 | 43 | 47
Completed | 34 | 27 | 35
Not Completed | 11 | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference Drug | Test Drug | Control | Total
Number analyzed (Participants) | 45 | 43 | 47 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 47 | 126
  >=65 years | 5 | 4 | 0 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (15.9) | 44.2 (14.5) | 43.1 (10.8) | 44.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 12 | 31
  Male | 35 | 34 | 35 | 104
Region of Enrollment [Number; unit: participants]
  United States | 45 | 43 | 47 | 135
Weight [Mean (Standard Deviation); unit: lbs] | 194.4 (45.49) | 199.5 (56.06) | 207.0 (49.75) | 200.4 (50.42)

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure Rate: Interdigital Disease
Description: A negative KOH and negative culture and no evidence of clinical disease as indicated by scores of 0 for each sign and symptom at Day 43.
Time Frame: Day 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 32 | 27 | 28
Participants | 9 | 9 | 1

2. Secondary Outcome: Effective Treatment: Interdigital Disease
Description: Negative KOH, negative fungal culture, no or mild (a score of 0 or 1) erythema and/or scaling with all other signs or symptoms being absent (score = 0) at Day 43 (Week6).
Time Frame: 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 32 | 27 | 28
Participants | 21 | 16 | 1

3. Primary Outcome: Complete Cure Rate: Moccasin Disease
Description: as for outcome 1
Time Frame: 43 Days
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 10 | 10 | 19
Participants | 2 | 0 | 0

4. Secondary Outcome: Effective Treatment: Mocassin Disease
Description: as for outcome 2
Time Frame: 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 10 | 10 | 19
Participants | 3 | 4 | 0

5. Secondary Outcome: Mycological Cure: Interdigital Disease
Description: Negative KOH and negative fungal culture at Day 43
Time Frame: 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 32 | 27 | 28
Participants | 27 | 20 | 4

6. Secondary Outcome: Mycological Cure: Mocassin Disease
Description: Negative KOH and negative fungal culture at Day 43
Time Frame: 43
Population: MITT
Measure: Number; unit: Participants
Arm/Group | Reference Drug | Test Drug | Control
Number analyzed (Participants) | 10 | 10 | 19
Participants | 5 | 5 | 1

ADVERSE EVENTS:
Arm/Group | Reference Drug | Test Drug | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43 | 0/47
Other Adverse Events (participants affected / at risk) | 10/45 | 10/43 | 7/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Drug (N=45) | Test Drug (N=43) | Control (N=47)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth Abcess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glucose Urine Present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other